CLINICAL TRIAL: NCT05805202
Title: Functional Implications of Rare Gene Mutations in aHUS Open the Door to Personalized Therapy
Acronym: aHUS-iPSC-EC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: aHUS-iPSC-EC
Record Dates: First submitted 2023-03-28; First posted 2023-04-07 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Atypical Hemolytic Uremic Syndrome
Keywords: Atypical hemolytic uremic syndrome; Induced pluripotent stem cells; Endothelial cells; Alternative complement pathway; Eculizumab; Drug screening (in vitro)
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome | interventions — Blood Specimen Collection; Urinalysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- aHUS Patient (Experimental): The study will include 110 patients consenting adult and pediatric patients with a diagnosis of atypical hemolytic uremic syndrome and carrying mutations in the MCP or DGKE genes. New patients will be selected through clinical and genetic screening of the inhabitants of a small island of South Italy (Linosa) with high incidence of patients affected by DGKE mutations and characterized by a high rate of endogamy
  Interventions: Other: Blood sampling and urine analysis
- Healthy volunteer (Other): 2 healthy subjects will undergo urine analysis (multistick) and only subjects with normal parameters will be enrolled as controls.
  Interventions: Other: Blood sampling and urine analysis

INTERVENTIONS:
Other: Blood sampling and urine analysis — A blood sample of 10- 20 ml from pediatric patients, 30-50 ml from adult patients will be collected for each patient and healthy voluntarees

SUMMARY:
Hemolytic Uremic Syndrome (HUS) is a rare disease characterized by rupture of red blood cells (hemolytic anemia), low platelet count (thrombocytopenia), and thrombotic occlusion of small vessels (thrombotic microangiopathy), with prevalent involvement of the kidneys.

SEU, in its typical form is caused by gastrointestinal infection with Escherichia coli.

The atypical form of SEU (aSEU), which is not caused by an Escherichia coli infection, is a very rare disease that may have a genetic origin; it affects both children and adults and may occur in a sporadic or familial form. Many studies have shown that about 60% of cases of atypical HUS are associated with genetic abnormalities of the complement system (particularly the so-called "alternative pathway"), which is a key part of the immune system for responding to infection. Complement consists of a series of proteins that, when activated, create a so-called "cascade," which leads to the elimination of the infectious agent, either directly or through other cells. Complement is finely regulated in such a way as to prevent damage to healthy cells in one's own body. Genetic defects in some of these complement regulatory proteins cause reduced protection of the endothelial surface (thus the vessel wall) against complement activation.

Recently, new mutations have been described in a gene unrelated to the complement pathway, the DKGE gene, which codes for the intracellular isoform of diacylglycerol kinase . In these patients, small renal vessel occlusion appears to occur as a result of altered endothelial cell proliferation and angiogenesis through mechanisms apparently unrelated to complement activation. However, to date these mechanisms are poorly studied. Throughout the entire project statistical methods will be applied to optimize the characterization of the abnormalities in phenotype and function of iPSC-EC derived from aHUS patients with either DGKE or MCP genetic abnormalities as compared with control iPSC-EC, including identifying potential drugs that could correct the abnormalities

ELIGIBILITY:
Inclusion Criteria:

* Adults and children with aHUS defined by history of microangiopathic hemolytic anemia and thrombocytopenia (hematocrit (Ht) <30%, hemoglobin (Hb) <10 g/dL, LDH >500 IU/L, undetectable haptoglobin, fragmented erythrocytes in the peripheral blood smear with negative Coomb's test, and platelet count <150,000/microL), associated with acute renal failure.
* Written informed consent

Exclusion Criteria:

* TTP (ADAMTS13 activity <10%)
* STEC-HUS (presence of stx and eae genes or Shiga-toxin in the stools and/or serum antibodies against Shiga-toxin and/or STEC LPS).
* Disseminated intravascular coagulation (prolonged thromboplastin time and lower than normal fibrinogen levels).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Generation and characterization of patient-specific and healthy donor iPSC | once during the study
Differentiation of iPSC into endothelial cells | once during the study
Characterizationof iPSC into endothelial cells | once during the study
Cell culture viability | once during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Centro di Ricerche Cliniche per le Malattie Rare "Aldo e Cele Daccò", Ranica, BG, Italy

IPD SHARING:
Plan to Share IPD: No